CLINICAL TRIAL: NCT04061213
Title: ATTR Amyloidosis in Elderly Patients With Aortic Stenosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 4083 / KEK-Nr. 2019-00880
Record Dates: First submitted 2019-08-15; First posted 2019-08-19 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Aortic Stenosis Symptomatic; Amyloidosis Cardiac
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with symptomatic severe aortic stenosis: Elderly patients referred for TAVR evaluation
  Interventions: Diagnostic Test: Tc-99m-DPD scintigraphy

INTERVENTIONS:
Diagnostic Test: Tc-99m-DPD scintigraphy — Myocardial scintigraphy

SUMMARY:
Severe aortic stenosis is defined with a mean transvalvular pressure gradient (MTPG) > 40mmHg and a calculated aortic valve area of < 1cm2. However, a considerable proportion of patients do have a MTPG < 40mmHg due to a reduced stroke volume (stroke volume indexed to body surface area ≤ 35ml/m2) despite a normal left ventricular ejection fraction (LVEF > 50%). This entity is termed paradoxical low flow low gradient aortic stenosis (PLFLG AS) and is associated with a worse prognosis.

ATTR amyloidosis is a disease of the elderly and might coexist in patients with severe aortic stenosis. Case reports and small observational studies suggest that senile ATTR amyloidosis could be frequent but underdiagnosed in patients with aortic stenosis. There is significant overlap between PLFLG AS and cardiac amyloidosis with regard to symptoms, increasing prevalence with age, concentric hypertrophy, impaired diastolic filling of the left ventricle (LV), as well as longitudinal LV dysfunction despite preserved ejection fraction - all features, which lead to a reduction in stroke volume, the underlying mechanism of the low flow condition as observed in PLFLG AS patients.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic, severe aortic stenosis

Exclusion Criteria:

* More than mild valvular disease of any other valve
* Other severe disease with a life expectancy < 1 year
* Participating in trial interfering with routine clinical practice or use of a non-CE marked device

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with symptomatic, severe aortic stenosis undergoing pre-evaluation for (transcatheter) aortic valve replacement
Sampling Method: Non-Probability Sample
Enrollment: 489 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with grade 2 or 3 cardiac uptake in scintigraphy and without pathological light chains in immunological assays | In-Hospital [7 days]
  Evaluation of incidence rate

SECONDARY OUTCOMES:
All-cause and cardiovascular mortality | 30 days, 12months
  Clinical Endpoints
CPET - maximal exercise capacity | In-Hospital [7 days]
  Functional Endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Stortecky, MD, Principal Investigator — Swiss Cardiovascular Center Bern
Locations (1):
- University Hospital Bern - Inselspital, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bernhard B, Leib Z, Dobner S, Demirel C, Caobelli F, Rominger A, Schutze J, Grogg H, Alwan L, Spano G, Boscolo Berto M, Lanz J, Pilgrim T, Windecker S, Stortecky S, Grani C. Routine 4D Cardiac CT to Identify Concomitant Transthyretin Amyloid Cardiomyopathy in Older Adults with Severe Aortic Stenosis. Radiology. 2023 Dec;309(3):e230425. doi: 10.1148/radiol.230425. PMID 38085082
- [Derived] Dobner S, Pilgrim T, Hagemeyer D, Heg D, Lanz J, Reusser N, Grani C, Afshar-Oromieh A, Rominger A, Langhammer B, Reineke D, Windecker S, Stortecky S. Amyloid Transthyretin Cardiomyopathy in Elderly Patients With Aortic Stenosis Undergoing Transcatheter Aortic Valve Implantation. J Am Heart Assoc. 2023 Aug 15;12(16):e030271. doi: 10.1161/JAHA.123.030271. Epub 2023 Aug 10. PMID 37581394